CLINICAL TRIAL: NCT04104204
Title: The Efficacy of Pain Control After Total Hip Replacement Between Ultrasound Guide Supra-inguinal Fascia Iliaca Block and Intrathecal Morphine: A Randomized Controlled Trial
Brief Title: The Efficacy of Pain Control After Total Hip Replacement Between Ultrasound Guided Supra-inguinal Fascia Iliaca Block and Intrathecal Morphine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Si 404/2019
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Total Hip Replacement; Ultrasound Guided Supra-inguinal Fascia Iliaca Block; Intrathecal Morphine; Postoperative Pain
Keywords: Total hip replacement; Ultrasound guided supra-inguinal fascia iliaca block; Intrathecal morphine; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine (Sham Comparator): Intrathecal morphine 0.1 mg, A sham subcutaneous injection of 0.5 ml normal saline at inguinal area
  Interventions: Drug: Intrathecal morphine
- Ultrasound guided supra-inguinal fascia iliaca block (Experimental): 0.25% bupivacaine 40 ml
  Interventions: Drug: Ultrasound guided supra-inguinal fascia iliaca block

INTERVENTIONS:
Drug: Intrathecal morphine — 0.5% Iso/Hyperbaric bupivacaine 2-3 ml add morphine 0.1 mg for spinal anesthesia
  Arms: Intrathecal morphine
Drug: Ultrasound guided supra-inguinal fascia iliaca block — Ultrasound guided supra-inguinal fascia iliaca block with 0.25% bupivacaine 40 ml and 0.5% Iso/Hyperbaric bupivacaine 2-3 ml without spinal morphine for spinal anesthesia
  Arms: Ultrasound guided supra-inguinal fascia iliaca block

SUMMARY:
Total hip replacement is one of major orthopedic surgery which result in severe postoperative pain especially at first 24 hours. Ultrasound guided regional anesthesia has become a part of multimodal analgesia.Ultrasound guided supra-inguinal fascia iliaca block is a new technique which can consistently cover femoral and lateral femoral cutaneous nerve. And with large volume (40ml), it may cover obturator nerve. This technique already proved to be useful for acute pain control in hip fracture or postoperative control in dynamic hip screw or nail insertion operation. However, it has not been compared with intrathecal morphine for total hip replacement yet.

DETAILED DESCRIPTION:
By using combine ultrasound guided supra-inguinal fascia iliaca block with periarticular infiltration with mutimodal analgesic drugs will have longer duration time to first rescue analgesic drug compared with combine intrathecal morphine with periarticular infiltration with multimodal analgesic drugs.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery of primary total hip replacement, body weight ≥40kg and BMI ≤35 kg/m2, competence to consent

Exclusion Criteria:

* contraindication to regional anesthesia, allergy to study drugs, skin infection at supra-inguinal fascia iliaca injection point, neurological deficit affecting the lower extremities, inability to use patient-controlled analgesia, GFR <50 mL/min

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic request (PCA fentanyl) | 48 hours
  Whether ultrasound guided supra-inguinal fascia iliaca block can increase pain free period of patients undergo total hip replacement under spinal block compare with intrathecal morphine or not

SECONDARY OUTCOMES:
Pain score | 48 hours
  Pain score at rest and on movement rating by numerical rating scale in 48-hr postoperative
Amount of rescue analgesic drugs | 48 hours
  Amount of PCA fentanyl

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Pangthipampai, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No